CLINICAL TRIAL: NCT04506060
Title: Evaluation of Renal Pretransplant Serology for BK Virus on the Risk of Post-transplant Viral Reactivation
Acronym: BKSEREIN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2020_843_0101
Record Dates: First submitted 2020-08-06; First posted 2020-08-10 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: BK Virus Nephropathy; Risk Factor; Kidney Transplantation
Keywords: BK Virus Nephropathy; risk factor; kidney transplantation; viral serology

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum of the transplant patient. In the transplanted patient, the search for the BK virus is traditionally carried out during visits in the first year after transplantation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: serum withdrawal — Serum of the transplant patient. In the transplanted patient, the search for the BK virus is traditionally carried out during visits in the first year after transplantation.

SUMMARY:
Due to the increasing importance of BKV infection on the survival of kidney transplants, a better knowledge, in the pretransplant phase, of the risk factors leading to viral reactivation could allow the follow-up physician to be more vigilant and better prevent this pathology. There are no commercial tests for BKV serology. In the virology laboratory, the investigators have developed the technique for producing "Virus-like particles" (VLP) that mimics the antigenic structure of the BK virus. The investigators plan to evaluate seroreactivity to the five BK virus serotypes in the recipient of a kidney transplant as a pretransplant and to compare this data with the detection or not of viral reactivation in the recipient during the first post-transplant year.

ELIGIBILITY:
Inclusion Criteria:

* adult kidney transplanted patients
* Renal transplant patients with regular virological follow-up (blood and urine for BKV) during the first year after transplantation.

Exclusion Criteria:

* Renal transplant patients with no follow-up for one year after transplantation (transplant failure, return to dialysis, death, follow-up outside the transplant centre)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Renal transplant patients with regular virological follow-up (blood and urine for BKV) during the first year after transplantation
Sampling Method: Non-Probability Sample
Enrollment: 378 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Serum antibody titre limit measurement of the five BK virus serotypes in pre-transplant patient | one year
  Serum antibody titre limit measurement of the five BK virus serotypes in pre-transplant patient. Optical density of serum antibody titer will be obtained by Elisa.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No